CLINICAL TRIAL: NCT06354829
Title: Creation of a Collection of Medical Images to Facilitate Their Use for Future Not-for-profit Research
Brief Title: Medical Images Collection Research
Acronym: MEDICALBUM
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MEDICALBUM
Record Dates: First submitted 2024-03-15; First posted 2024-04-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Kidney Diseases; Brain Diseases
Keywords: Medical images; Repository; Kidney diseases; Cerebral diseases; Database
MeSH Terms: conditions — Kidney Diseases; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney cohort: Once assigned to the renal cohort, the relevant set of images will then be further assigned to a specific subpopulation depending on the pathology. In parallel, the associated anamnestic, demographic, and clinical data, will be included in a purpose-designed electronic Case Report Form (eCRF).
  Interventions: Diagnostic Test: Medical imaging procedures
- Cerebral cohort: Once assigned to the cerebral cohort, the relevant set of images will then be further assigned to a specific subpopulation depending on the pathology. In parallel, the associated anamnestic, demographic, and clinical data, will be included in a purpose-designed eCRF.
  Interventions: Diagnostic Test: Medical imaging procedures

INTERVENTIONS:
Diagnostic Test: Medical imaging procedures — The following medical imaging procedure will b applied: Magnetic resonance images (MRI), computerized tomography images (CT), and ultrasound images (US).

SUMMARY:
This is a not-for-profit project for the collection, archiving and reuse of magnetic resonance imaging, computed tomography and ultrasound images, and related demographic and clinical data, for research purposes only.

DETAILED DESCRIPTION:
The collection of medical images and related data will be proposed to each participant to concluded or ongoing clinical trials promoted or partnered by the Mario Negri Institute for Pharmacological Research (IRFMN) requiring the collection of images or subject who perform a clinical practice examination at the Hospitals that adopted the image acquisition protocols of IRFMN. Each subject will be provided with an informed sheet and will be asked to provide consent to donate his/her medical images and related data for future research. For participants in new clinical trials, the consent sheet of the study will be accompanied by this trial's consent sheet.

In addition to the information reported in the specific trial information sheet, each subject shall have access to the list of studies included in the Clinical Trials Register of IRFMN/Bioengineering Department that are reusing their medical image data.

Any new study protocol promoted by IRFMN and which provides for the use of medical images stored in this trial will be submitted to the local Ethics Committee for approval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: Adults ≥ 18 years; Subjects with no previous history of kidney or cerebral disease
* Patients: Adults ≥ 18 years; Subjects with renal or cerebral disease

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants to concluded or ongoing clinical trials promoted or partnered by IRFMN requiring the collection of images or subjects who perform a clinical practice examination at the Hospitals that adopted the image acquisition protocols of IRFMN.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2049-09 (Estimated); Study Completion 2049-09 (Estimated)

PRIMARY OUTCOMES:
Creation of a medical images collection | Image acquisitions at baseline
  Collection of medical images and related data of participants to concluded or ongoing clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Matias Trillini, PhD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Center for Rare Disease Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caroli A, Antiga L, Conti S, Sonzogni A, Fasolini G, Ondei P, Perico N, Remuzzi G, Remuzzi A. Intermediate volume on computed tomography imaging defines a fibrotic compartment that predicts glomerular filtration rate decline in autosomal dominant polycystic kidney disease patients. Am J Pathol. 2011 Aug;179(2):619-27. doi: 10.1016/j.ajpath.2011.04.036. Epub 2011 Jun 17. PMID 21683674
- [Background] Caroli A, Capelli S, Napolitano A, Cabrini G, Arrigoni A, Pezzetti G, Previtali M, Longhi LG, Zangari R, Lorini FL, Sessa M, Remuzzi A, Gerevini S. Brain diffusion alterations in patients with COVID-19 pathology and neurological manifestations. Neuroimage Clin. 2023;37:103338. doi: 10.1016/j.nicl.2023.103338. Epub 2023 Jan 28. PMID 36731251
- [Background] Soliveri L, Bozzetto M, Brambilla P, Caroli A, Remuzzi A. Hemodynamics in AVF over time: A protective role of vascular remodeling toward flow stabilization. Int J Artif Organs. 2023 Oct-Nov;46(10-11):547-554. doi: 10.1177/03913988231191960. Epub 2023 Sep 27. PMID 37753863
- [Background] Villa G, Daina E, Brambilla P, Gamba S, Leone VF, Carrara C, Rizzo P, Noris M, Remuzzi G, Remuzzi A, Caroli A. Functional Magnetic Resonance Imaging to Monitor Disease Progression: A Prospective Study in Patients with Primary Membranoproliferative Glomerulonephritis. Nephron. 2024;148(6):367-378. doi: 10.1159/000534893. Epub 2023 Nov 3. PMID 37926085